CLINICAL TRIAL: NCT04863092
Title: Intervention to Educate and Improve Underrepresented Populations' Participation in Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-0590.cc; P30CA046934 (NIH)
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: It uses a pre- and post-design to evaluate participants' changes in knowledge of and intentions to in CTs by comparing outcomes at baseline to outcomes after exposure to the CHE educational intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Underrepresented Population (Experimental): A primary emphasis is placed on those from underrepresented populations, including Hispanics, residents of outlying rural areas, and those in areas of poverty
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — The workshops will last approximately 60 minutes, with 20 minutes to educate participants and 10 minutes to discuss the materials and answer any questions. Prior to and after the presentation, the CHE will administer the pre- and post-intervention survey to participants. Group sizes will be capped to 25 individuals per group.

SUMMARY:
This proposal aims to leverage ongoing community outreach efforts and the Cancer Center's aims to improve recruitment to clinical trials by educating the catchment and making referrals to engage current UCCC patients not taking advantage of available CTs at this institution and affiliated hospitals. The Cancer Prevention and Control Program within UCCC works to develop and evaluate novel approaches to primary prevention, disseminate preventative interventions in population-based settings, and to improve health services delivery and outcomes for cancer patients and survivors. A primary emphasis is placed on those from underrepresented populations, including Hispanics, residents of outlying rural areas, and those in areas of poverty. Efforts to meet the Cancer Center's priorities include interventions to promote awareness and recruitment of eligible patients to available CTs in the catchment area (the state of Colorado).

DETAILED DESCRIPTION:
Clinical Trial Education Intervention: The educational intervention will be delivered to approximately 200 participants by the Community Health Educators (CHEs) who will conduct workshops to deliver content and educational materials to patients about the importance of participating in cancer clinical trials. The workshops will last approximately 60 minutes, with 20 minutes to educate participants and 10 minutes to discuss the materials and answer any questions. Prior to and after the presentation, the CHE will administer the pre- and post-intervention survey to participants. Group sizes will be capped to 25 individuals per group.

Additionally, the CHE and/or Patient Navigators (PNs) will set up pathways for communication with key personnel (i.e. nurse navigators, clinical research coordinators, investigators) from partnering hospitals and clinics to facilitate patient referrals and evaluation for eligibility for clinical trials. The CHE and/or PN will keep track of those individuals that are referred by the partner hospital and clinics to track if the PN referral resulted in enrollment and participation in a clinical trial. The CHE and/or PN will also record and report quarterly the number of: (a) persons referred to therapeutic/intervention CTs at the UCCC and partnering hospitals; (b) referred persons screened for therapeutic/intervention CTs at the UCCC and partnering hospitals; (c)referred persons enrolled in therapeutic/ intervention CTs at the UCCC and partnering hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be over 18 years old
4. English and/or Spanish Speaking

Exclusion Criteria:

1. Individuals who do not meet eligibility criteria, including individuals who do not speak English or Spanish [at the discretion of the CHE or PN upon recruitment];
2. Decisionally-challenged adults with cognitive or personality impairment or due to intoxication (alcohol or drugs) that might interfere with their ability to consent or participate in the study [at the discretion of the CHE or PN upon recruitment];
3. Individuals from vulnerable populations (e.g., inmates, homeless, pregnant women, and those with auditory impairment [at the discretion of the CHE or PN upon recruitment].
4. Individuals under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Change in knowledge and understanding of and intent to participate in Clinical Trials (CTs) | 36 months
  Using questionnaires to measure the change in knowledge of and understanding and intent to participate in CTs
Number of patients referred, screened, and enrolled into cancer related therapeutic CTs | 36 months
  Monitoring the number of referrals to and enrollment in CTs will help determine effectiveness of educational materials.

SECONDARY OUTCOMES:
Change in number of underrepresented patients participating in cancer related therapeutic CTs | 36 months
  In collaboration with the Cancer Clinical Trials Office (CCTO), the investigators will obtain quarterly demographic data for all participants across all clinical trials within the system and affiliate hospitals
Identify relationships between sociodemographic variables and the attitudes towards CTs | 36 months
  For future studies, this can help provide insight as to what sociodemographic variables to target to increase CTs enrollment in the catchment area

OTHER OUTCOMES:
PN-referred persons screened for cancer related therapeutic CTS; | 36 months
  The number of patients who interact with the site and connect with the PN for other services.
PN-referred persons enrolled in related therapeutic CTS; | 36 months
  The number of patients who interact with the site and connect with the PN for other services.
connected to care services such as health insurance, treatment assistance programs | 36 months
  The number of patients who interact with the site and connect with the PN for other services.
facilitate other services such as language translation, appointment scheduling, transportation, and childcare. | 36 months
  The number of patients who interact with the site and connect with the PN for other services.

CONTACTS AND LOCATIONS:
Overall Officials: Evelinn Borrayo, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No